CLINICAL TRIAL: NCT01799798
Title: TRANSLATIONAL THERAPY IN PATIENTS WITH OSTEOGENESIS IMPERFECTA - A PILOT TRIAL ON TREATMENT WITH THE RANKL-ANTIBODY DENOSUMAB
Acronym: OI-AK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. med. Joerg Oliver Semler, Head of the outpatient center for sceletal dysplasias, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-1574
Record Dates: First submitted 2013-02-14; First posted 2013-02-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Osteogenesis Imperfecta
Keywords: Osteogenesis imperfecta; COL1A1/A2; Denosumab; Bisphosphonates; Children; Areal bone mineral density
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Denosumab subcutaneously (Experimental)
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Denosumab will be given subcutaneously in a dosage of 1mg/kg body weight every 12 weeks. 4 interventions are planned until trial week 36. There is no control group planned.

SUMMARY:
Pilot study to assess the efficacy of a therapy with the RANKL-antibody denosumab in children 5-10 years of age with mutation in COL1A1 or COL1A2 leading to Osteogenesis imperfecta. Efficacy will be assessed by DXA measurements at the lumbar spine of the areal bone mineral density (BMD) which is the most frequently used parameter in trials investigating osteoporosis.

The hypothesis of the study is:

Osteoclastic activity which is increased in OI could be reduced by inhibition of osteoclast maturation. Denosumab inhibits maturation of the osteoclasts by inhibiting RANKL. BMD could be increased during a 36 week treatment course with denosumab measured after 48 weeks.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects between 5 years and 10 years of age with molecular proven Osteogenesis imperfecta (COL1A1/A2 mutation)
* Subjects must have been treated for a minimum of 2 years with bisphosphonates prior to study entry

Exclusion Criteria:

* Hypocalcemia (<1.03 mmol/l ionized Calcium)
* Subjects with reduced renal function (estimated GFR (Schwartz formula) <30ml/min/1.73m2)
* Any other abnormal finding such as physical examination or laboratory evaluation, in the opinion of the investigator that is indicative of a disease that would compromise the safety of the patient when getting denosumab s.c.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Changes of bone mineral density (BMD [g/cm2]) in lumbar spine after 36 weeks of treatment with denosumab. Changes will be calculated between baseline and study week 48. | 48 weeks

SECONDARY OUTCOMES:
Decrease of osteoclastic activity measured by urinary deoxypyridinoline (DPD). | 14 days (DPD)
Parathormone in study week 12, 24, 36 and 48 compared to baseline. | 12 weeks
  Descriptive statistical analysis
N-Telopeptides in study week 12, 24, 36 and 48 compared to baseline. | 12 weeks
  descriptive statistical analysis
Osteocalcin in study week 12, 24, 36 and 48. | 12 weeks
  descriptive statistical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Oliver Semler, MD, Principal Investigator — University Cologne, Childrens Hospital, Cologne, Germany
Locations (1):
- University Cologne, Childrens Hospital, Cologne, Germany, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Semler O, Netzer C, Hoyer-Kuhn H, Becker J, Eysel P, Schoenau E. First use of the RANKL antibody denosumab in osteogenesis imperfecta type VI. J Musculoskelet Neuronal Interact. 2012 Sep;12(3):183-8. PMID 22947550